CLINICAL TRIAL: NCT02385019
Title: A Phase 1/2 Trial of Donor Regulatory T-cells for Steroid-Refractory Chronic Graft-versus-Host-Disease
Acronym: TREGeneration
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Medicina Molecular João Lobo Antunes (Other)
Collaborators: Hospital de Santa Maria, Portugal (Other); IPOFG Lisboa, Portugal (Unknown); IPOFG Porto, Portugal (Unknown)
Responsible Party: Principal Investigator, Joao F. Lacerda, MD PhD, Associate Professor of Medicine, Instituto de Medicina Molecular João Lobo Antunes
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREGeneration-Portugal
Record Dates: First submitted 2015-03-01; First posted 2015-03-11 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Graft vs Host Disease
Keywords: Allogeneic hematopoietic stem cell transplantation; Graft vs host disease; Regulatory T cells
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Administration of 0.5 x 10ˆ6 donor Treg/kg (Experimental): First group of 5 patients will receive a total of 0.5 x 10ˆ6 donor Treg/kg. Part of Phase 1 study.
  Interventions: Biological: Donor regulatory T cell adoptive immunotherapy in chronic graft versus host disease
- Administration of 1.0 x 10ˆ6 donor Treg/kg (Experimental): Second group of 5 patients will receive a total of 1.0 x 10ˆ6 donor Treg/kg. Part of Phase 1 study.
  Interventions: Biological: Donor regulatory T cell adoptive immunotherapy in chronic graft versus host disease
- Administration of 2.0-3.0 x 10ˆ6 donor Treg/kg (Experimental): Third group of 5 patients will receive a total of 2.0-3.0 x 10ˆ6 donor Treg/kg. Part of Phase 1 study.
  Interventions: Biological: Donor regulatory T cell adoptive immunotherapy in chronic graft versus host disease
- Administration of MTD of donor T reg (Experimental): Preliminary Phase 2 study will include another 5 to 10 patients at the MTD identified in the Phase 1 study
  Interventions: Biological: Donor regulatory T cell adoptive immunotherapy in chronic graft versus host disease

INTERVENTIONS:
Biological: Donor regulatory T cell adoptive immunotherapy in chronic graft versus host disease — Regulatory T cells selected by a sequential 2 step procedure:
  1. - Negative selection of CD8 and CD19 cells
  2. - Positive selection of CD25 cells

SUMMARY:
Phase 1/2 clinical study for the treatment of steroid-refractory chronic graft versus host disease after an allogeneic transplant of hematopoietic progenitors with donor CliniMACS-selected regulatory T cells

DETAILED DESCRIPTION:
Phase 1/2 clinical study evaluating safety (Phase 1) and preliminary efficacy (Phase 2) of donor regulatory T cells for patients with steroid-refractory chronic graft versus host disease (GVHD) after allogeneic hematopoietic stem cell transplantation (HSCT).

Patients must have persistent signs and symptoms despite the use of prednisone or equivalent at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day), for at least 4 weeks without complete resolution of signs and symptoms. Occasional patients requiring lower doses of prednisone will be eligible if associated with other immunosuppressive drugs.

Phase 1 clinical trial will include groups of 5 patients sequentially treated with: 0.5 x 10ˆ6, 1.0 x 10ˆ6, 2-3 x 10ˆ6 donor Treg/kg. Phase 2 clinical trial will include another 5 to 10 patients treated with MTD.

Donor Treg will be selected by the following sequential steps:

1. - negative depletion of CD8 and CD19 cells
2. - positive selection of CD25 cells

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have persistent signs and symptoms despite the use of prednisone or equivalent at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day), for at least 4 weeks without complete resolution of signs and symptoms. Occasional patients requiring lower doses of prednisone will be eligible if associated with other immunosuppressive drugs.
2. Stable immunosuppressive medication in the 4 weeks prior to initiation of treatment
3. PS 0-2 ECOG
4. Adequate liver, kidney, lung and hematopoietic system functions

Exclusion Criteria:

1. Pediatric patients
2. Pregnant women
3. Ongoing prednisone requirement >1 mg/kg/day (or equivalent)
4. Concurrent use of calcineurin-inhibitor plus sirolimus (either agent alone is acceptable)
5. New immunosuppressive medication in the 4 weeks prior
6. Extra-corporeal Photopheresis or rituximab therapy in the 4 weeks prior
7. Exposure to T-cell or IL-2 targeted medication (e.g. ATG, alemtuzumab, basiliximab, denileukin diftitox) within 100 days prior
8. Donor lymphocyte infusion within 100 days prior
9. Active malignant relapse
10. Active uncontrolled infection
11. HIV-infected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression of graft versus host disease according to the 2014 NIH consensus criteria and myelosuppression after the administration of 3 doses of donor regulatory T cells / kg recipient's body weight: 0.5 x 10ˆ6, 1.0 x 10ˆ6 and 2.0-3.0 x 10ˆ6 cells | Response evaluated 12 weeks after infusion
  Progression of graft versus host disease and myelosuppression are indicators of toxicity and MTD associated with the infusion of donor regulatory T cells

SECONDARY OUTCOMES:
Chronic graft versus host disease improvement according to the 2014 NIH consensus criteria following the infusion of donor regulatory T cells | Response evaluated 12 weeks after infusion
Total lymphocyte, CD4, CD8 and regulatory T cell counts after the infusion of donor regulatory T cells for the treatment of chronic graft versus host disease | Response evaluated 12 weeks after infusion
Survival at 1 year after administration of donor regulatory T cells in patients with chronic graft versus host disease | Response evaluated 12 months after infusion

CONTACTS AND LOCATIONS:
Locations (3):
- Portugal (3):
  - Instituto Portugues de Oncologia, Lisbon
  - Hospital de Santa Maria, Faculdade de Medicina da Universidade de Lisboa, Instituto de Medicina Molecular, Lisbon
  - Instituto Portugues de Oncologia, Porto

REFERENCES:
- [Derived] Soares MV, Escamilla Gomez V, Azevedo RI, Pereira PNG, Caballero-Velazquez T, Mendes L, Alho AC, Garcia-Guerrero E, Garcia-Calderon CB, Tharmaratnam K, Cabral IA, Ribeiro AC, Juncal C, Roncon S, Pais AT, Rodriguez-Gil A, Espada ELDS, Rodrigues A, Garcao A, Yaspo ML, Warnatz HJ, Lehrach HR, Ward L, Barbosa-Morais NL, Quintas AM, Palmela P Sr, Caldas CMF, Ferreira R, Leite L, Martins C, Lourenco F, Moreno R, Campilho F, Cheyne CP, Garcia-Finana M, Campos AM, Baron F, Arpinati M, Hoffmann P, Edinger M, Koreth J, Ritz J, Pinho Vaz C, Perez-Simon JAA, Lacerda JF. Phase I/II Trials of Donor Regulatory T Cells for the Treatment of Steroid-Refractory Chronic Graft versus Host Disease. Blood Adv. 2026 Feb 4:bloodadvances.2025017996. doi: 10.1182/bloodadvances.2025017996. Online ahead of print. PMID 41637631